CLINICAL TRIAL: NCT04831671
Title: A Pilot Randomised Prospective Comparison of Two Approaches for Tibial Nailing Using Clinical and Novel Imaging Outcome Measures
Brief Title: MRI Assessment of Cartilage Damage in Tibial Nailing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mr Andrew Carrothers, Consultant Trauma and Orthopaedic Surgeon, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A095899
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Tibial Fractures
Keywords: MRI; Cartilage Damage; Surgical Techniques
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Masking Description: It is not possible to mask participants or investigators as the surgical interventions in each arm will have different scars, making blinding impossible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infra-patella nailing (Active Comparator): Participants will have their closed tibial shaft fracture treated with an intra-medullary nail inserted through an infra-patella approach.
  Interventions: Other: Surgical Approach - Infra-patella nailing
- Supra-patella nailing (Experimental): Participants will have their closed tibial shaft fracture treated with an intra-medullary nail inserted through an supra-patella approach.
  Interventions: Other: Surgical Approach - Supra-patella nailing

INTERVENTIONS:
Other: Surgical Approach - Infra-patella nailing — The intra-medullary nail will be introduced via an infra-patella incision.
  Arms: Infra-patella nailing
Other: Surgical Approach - Supra-patella nailing — The intra-medullary nail will be introduced via a supra-patella incision.
  Arms: Supra-patella nailing

SUMMARY:
Fractures of the tibia (shin bone) are frequently treated with a metal nail that is passed down the inside of the bone (an intra-medullary nail). This nail is inserted through the top of the tibia at the level of the knee joint. There are two ways for the nail to be inserted - either through an incision below the patella (kneecap) or above the patella.

The benefit of the incision above the patella is that it can make it technically easier to insert the nail into the correct position. However, the perceived risk of damage to the knee cartilage has prevented this technique from being widely adopted.

The investigators will use MRI scanning to assess the cartilage for damage using both techniques. The results will enable the investigators to determine if the theoretical risk of cartilage damage is found in real-world scenarios and to generate data for further, larger studies.

DETAILED DESCRIPTION:
Intra-medullary nailing is a common form of treatment for a variety of tibial shaft fractures. Traditionally this has been done via an infra-patella approach. More recently the use of a supra-patella approach has become more popular. However, there are concerns that the supra-patella approach may cause unacceptable damage to the cartilage of the patello-femoral joint (PFJ).

This study will use a novel MRI technique developed at the University of Cambridge to compare the amount of damage caused to the knee joint by both infra- and supra-patella nailing techniques. Specific cartilage assessment sequences will enable a fuller assessment of cartilage damage than can be achieved with normal structural sequences. Participants will also be asked to complete Patient Reported Outcome Measures (PROMs) regarding their injury to assess their clinical outcome.

Infra-patella and supra-patella nailing techniques are now both routine methods of carrying out intra-medullary nailing of the tibia. Further evidence is required, however, in order to fully assess whether one method is superior to the other.

ELIGIBILITY:
Inclusion Criteria:

* Closed tibial shaft fracture suitable for intramedullary nailing
* Able to consent
* Able to undergo MRI scanning
* Able to attend follow up for 6 months post operatively
* Suitable for surgery

Exclusion Criteria:

* Polytrauma
* Ipsilateral acute ligamentous knee injury
* A contra-indication to MRI scanning

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in cartilage appearance by MRI Assessment | Pre-intervention, Day 1 post operatively, 6 months
  Change in cartilage appearance of the ipsilateral knee using MRI scanning

SECONDARY OUTCOMES:
Change in Lysholm Knee Score | Pre-intervention, 6 weeks, 12 weeks, 6 months
  Change in Lysholm Knee Score (Scored 0-100, higher scores are better)
Change in Tegner Activity Scale | Pre-intervention, 6 weeks, 12 weeks, 6 months
  Change in Tegner Activity Scale (Scored 0-10, higher scores are move active)
Change in EQ-5D-5L | Pre-interventional , 6 weeks, 12 weeks, 6 months
  Change in EQ-5D-5L (EuroQol 5 Dimension 5 Level) (Each domain scored 1-5, lower scores are better)

OTHER OUTCOMES:
Bony Union of Fracture | 6 weeks
  Bony union will be assessed by plain radiograph
Bony Union of Fracture | 12 weeks
  Bony union will be assessed by plain radiograph
Bony Union of Fracture | 6 months
  Bony union will be assessed by plain radiograph
Post-operative Complications | up to 6 months
  Post operative complications will be recorded
Return to work/employment status | 6 months
  Patient return to normal activity will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Carrothers, FRCS (Tr & Orth), Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No